CLINICAL TRIAL: NCT03457805
Title: Prostatic Artery Embolization (PAE) in Patients With Advanced Prostate Cancer: A Pilot Study.
Brief Title: Prostatic Artery Embolization in Advanced Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dominik Abt (Other)
Responsible Party: Sponsor-Investigator, Dominik Abt, Dr. med., Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTU17/028
Record Dates: First submitted 2018-02-22; First posted 2018-03-08 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Prostate Cancer; Bladder Outlet Obstruction
Keywords: prostate cancer; prostate; embolization; minimally invasive; cytoreductive therapy
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neck Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostatic Artery Embolization (PAE) (Other): PAE performed under local anesthesia using officially approved microspheres.
  Interventions: Device: Prostatic Artery Embolization

INTERVENTIONS:
Device: Prostatic Artery Embolization — PAE is performed under local anesthesia using commercially available and approved microspheres (study is not limited to a specific manufacturer or product).

SUMMARY:
This is a pilot study assessing efficacy and safety in patients with advanced prostate cancer.

DETAILED DESCRIPTION:
PAE has been shown to be safe and effective in the treatment of prostatic bleeding and lower urinary tract symptoms arising from bladder outlet obstruction.

Advanced (defined as locally advanced, metastatic or both in this study) PCA is frequently associated with both of these conditions. The currently most frequently performed palliative surgical treatment is TURP. Though performed endoscopically, TURP is associated with significant side effects in this setting. PAE has been shown to have a superior side-effect profile in the treatment of bladder outlet obstruction compared to TURP.

In addition, there is growing evidence that patients with advanced PCA might benefit from cytoreductive therapy (e.g. radical prostatectomy or external beam radiation therapy). However, recent methods of cytoreductive treatment of PCA hold the risk of being highly invasive and are associated with severe side effects. PAE might represent a minimally invasive alternative in this setting.

Therefore, efficacy and safety of PAE in patients with advanced prostate cancer is assessed in this pilot-study.

ELIGIBILITY:
Inclusion Criteria

* Advanced PCA (i.e., locally advanced, metastatic, combination of both. This includes T3-4, any T in case of N1 and any T in case of M1a/b/c)
* PAE is indicated for the treatment of Lower urinary tract symptoms like bladder outlet obstruction or recurrent prostatic bleeding.
* IPSS at baseline ≥ 8
* Witten informed consent

Exclusion Criteria:

* Curative treatment of PCA intended
* Contraindications for MRI
* Renal impairment (GFR < 30ml/min)
* Allergy to i.v. contrast medium
* Vascular conditions that seem to make successful PAE impossible (e.g. severe atherosclerosis, severe tortuosity in the aortic bifurcation or internal iliac vessels)
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Drug-treatments for advanced prostate cancer (e.g., hormonal therapy or chemotherapy) established within 30 days prior to PAE.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-02 (Actual); Primary Completion 2021-07-02 (Estimated); Study Completion 2021-08-02 (Estimated)

PRIMARY OUTCOMES:
Reduction of Lower Urinary Tract Symptoms | Baseline and 12 weeks
  Change of total score of International Prostate Symptoms Score (IPSS; range 0 points (no symptoms) to 35 points (severe symptoms))

SECONDARY OUTCOMES:
Reduction of Lower Urinary Tract Symptoms | Baseline and 6 weeks
  Change of total score of International Prostate Symptoms Score (IPSS; range 0 points (no symptoms) to 35 points (severe symptoms))
Reduction of Lower Urinary Tract Symptoms | Baseline and 6 months
  Change of total score of International Prostate Symptoms Score (IPSS; range 0 points (no symptoms) to 35 points (severe symptoms))
Reduction of Lower Urinary Tract Symptoms | Baseline and 12 months
  Change of total score of International Prostate Symptoms Score (IPSS; range 0 points (no symptoms) to 35 points (severe symptoms))
Occurrence of macroscopic hematuria | From time of PAE to study completion (1 year)
  Assessment of occurrence of hematuria according to CTCAE v.4.03 classification
Reduction of Prostate symptoms | baseline and 6 weeks
  Change of CPSI total score (Chronic prostatitis symptoms score; range 0 points (no symptoms) to 43 points (severe symptoms))
Reduction of Prostate symptoms | baseline and 12 weeks
  Change of CPSI total score (Chronic prostatitis symptoms score; range 0 points (no symptoms) to 43 points (severe symptoms))
Reduction of Prostate symptoms | baseline and 6 months
  Change of CPSI total score (Chronic prostatitis symptoms score; range 0 points (no symptoms) to 43 points (severe symptoms))
Reduction of Prostate symptoms | baseline and 12 months
  Change of CPSI total score (Chronic prostatitis symptoms score; range 0 points (no symptoms) to 43 points (severe symptoms))
Occurrence of urinary incontinence | 6 week after PAE
  Assessment of ICS-SF questionnaire
Occurrence of urinary incontinence | 12 week after PAE
  Assessment of ICS-SF questionnaire
Occurrence of urinary incontinence | 6 months after PAE
  Assessment of ICS-SF questionnaire
Occurrence of urinary incontinence | 12 months after PAE
  Assessment of ICS-SF questionnaire
Changes of free urinary flow rate | Baseline and 6 weeks
  Measurement of urinary stream (mL/s) by urinary flow rate measurement
Changes of free urinary flow rate | Baseline and 12 weeks
  Measurement of urinary stream (mL/s) by urinary flow rate measurement
Changes of free urinary flow rate | Baseline and 6 months
  Measurement of urinary stream (mL/s) by urinary flow rate measurement
Changes of free urinary flow rate | Baseline and 12 months
  Measurement of urinary stream (mL/s) by urinary flow rate measurement
Changes of post void residual urine | Baseline and 6 weeks
  Measurement of post void residual urine (mL) by transabdominal ultrasound
Changes of post void residual urine | Baseline and 12 weeks
  Measurement of post void residual urine (mL) by transabdominal ultrasound
Changes of post void residual urine | Baseline and 6 months
  Measurement of post void residual urine (mL) by transabdominal ultrasound
Changes of post void residual urine | Baseline and 12 months
  Measurement of post void residual urine (mL) by transabdominal ultrasound
Rate of local reinterventions | During 1 year study period
  Assessment of number and type of reinterventions for prostate and bladder problems
Intraoperative Adverse Events | While PAE is performed (intra-operatively)
  Assessment of adverse events that are at least possibly related to study procedure according to Clavien-Dindo and CTCAE
Adverse Events | 6 weeks after PAE
  Assessment of adverse events that are at least possibly related to study procedure according to Clavien-Dindo and CTCAE
Adverse Events | 12 weeks after PAE
  Assessment of adverse events that are at least possibly related to study procedure according to Clavien-Dindo and CTCAE
Adverse Events | 6 months after PAE
  Assessment of adverse events that are at least possibly related to study procedure according to Clavien-Dindo and CTCAE
Adverse Events | 12 months after PAE
  Assessment of adverse events that are at least possibly related to study procedure according to Clavien-Dindo and CTCAE
Feasibility of PAE | While PAE is performed (intra-operatively)
  Possibility of successful completion of PAE in the study cohort defined by compete stasis of blood flow in the prostate
Estimation of tumor burden | Baseline and 24h after PAE
  Changes of Prostate Specific Antigen
Estimation of tumor burden | Baseline and 6 weeks after PAE
  Changes of Prostate Specific Antigen
Estimation of tumor burden | Baseline and 12 weeks after PAE
  Changes of Prostate Specific Antigen
Estimation of tumor burden | Baseline and 6 months after PAE
  Changes of Prostate Specific Antigen
Estimation of tumor burden | Baseline and 12 months after PAE
  Changes of Prostate Specific Antigen
Estimation of tumor volume | Baseline and 12 weeks after PAE
  Change of tumor volume calculated by magnetic resonance imaging
Prostate volume | Baseline and 12 weeks after PAE
  Change of prostate volume calculated by magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Abt, MD, Principal Investigator — St. Gallen Cantonal Hospital, Dept. of Urology, Rorschacherstrasse 95, 9007 St. Gallen
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Decision will be made individually up on request and based on approval by our local ethics committee.

REFERENCES:
- [Derived] Burkhardt O, Abt D, Hechelhammer L, Kim O, Omlin A, Schmid HP, Engeler D, Zumstein V, Mullhaupt G. Prostatic Artery Embolization in Patients with Advanced Prostate Cancer: A Prospective Single Center Pilot Study. Cardiovasc Intervent Radiol. 2024 Jun;47(6):771-782. doi: 10.1007/s00270-024-03679-z. Epub 2024 Feb 28. PMID 38416176